CLINICAL TRIAL: NCT00805753
Title: A Dose-Finding Pilot Study of ACTH on the Serum Lipoprotein Profile and Proteinuria in Patients With Idiopathic Membranous Nephropathy (MN)
Brief Title: Dose-Finding Pilot Study of ACTH in Patients With Idiopathic Membranous Nephropathy
Acronym: MN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Fernando Fervenza, M.D., Ph.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-006328
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 ACTH 40 units (Active Comparator): Receive ACTH at the dose of 40 units sub-cutaneously for up to 12 weeks. If at day 91 no response has been shown, you will have the option to increase the dose of ACTH to 80 units for up to an additional 120 days.
  Interventions: Drug: ACTH
- Arm 2 ACTH 80 units (Active Comparator): Receive ACTH at the dose of 80 units sub-cutaneously for up to 12 weeks.
  Interventions: Drug: ACTH

INTERVENTIONS:
Drug: ACTH — comparison of different dosages of drug
  Other Names: H.P. Acthar Gel

SUMMARY:
This pilot study is aimed at demonstrating the effectiveness of ACTH (H.P. Acthar Gel) on the lipid profile and proteinuria in participants with MN. ACTH or adrenocorticotrophin is a hormone produced by the pituitary gland (a gland at the base of your brain) that is involved in stimulating your adrenal glands to secrete a number of steroid products (e.g. cortisol, aldosterone, corticosterone, and others) that are important in keeping you alive. The drug used in this study has been approved by the Food and Drug Administration (FDA) for routine clinical use in the treatment of patients with proteinuria and patients with idiopathic nephrotic syndrome such as idiopathic MN. However, the most adequate dose to use has not been adequately assessed. This is the reason for conducting this research study.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic MN with diagnostic biopsy performed less than 36 months from the time of dose randomization.
2. Age > 18 years.
3. Patients need to be treated with an ACEI and/or ARB, for at least 3 months prior to ACTH treatment and have adequately controlled blood pressure
4. Proteinuria of >4.0 on a 24-hour urine collection.
5. Estimated GFR >40 ml/min/1.73m2 while taking ACEI/ARB therapy.

Exclusion Criteria:

1. Age <18 years.
2. Estimated GFR <40 ml/min/1.73m2, or serum creatinine >2.0 mg/dl.
3. Renal biopsy showing more than 30% glomerulosclerosis and/or tubular atrophy.
4. Patient must be off glucocorticoid, calcineurin inhibitors (cyclosporin A, tacrolimus) or mycophenolic mofetil for >1 month, and alkylating agents or rituximab for >6 months.
5. Resistance to the following immunosuppressive routines e.g. steroids alone, calcineurin inhibitors plus or minus steroids, cytotoxic agents plus or minus steroids.
6. Patients with active infections or secondary causes of MN.
7. Type 1 or 2 diabetes mellitus.
8. Pregnancy or nursing.
9. Acute renal vein thrombosis documented prior to entry by renal US or CT scan and requiring anticoagulation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in proteinuria | baseline, 3 months
Change in LDL cholesterol, HDL cholesterol, and triglycerides | baseline, 3 months
Change in side effects/toxicity | baseline, 3 months

SECONDARY OUTCOMES:
Number of subjects with CR or PR | 3 months
The effect of maximizing angiotensin II blockade on proteinuria | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C Fervenza, M.D., Ph.D, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952